CLINICAL TRIAL: NCT06993662
Title: The Effectiveness and Efficacy of the Combination of Pharmacotherapy and Cognitive Behavioral Psychotherapy Under the Recovery Perspective for Patients With Mental Health Disorders
Brief Title: The Combination of Pharmacotherapy and Cognitive Behavioral Psychotherapy Under the Recovery Perspective.
Acronym: RAKGEOCBT
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rakitzi, Stavroula (Other)
Responsible Party: Principal Investigator, Dr. Stavroula Rakitzi, Dr. phil., Dipl.-Psych., Clinical psychologist and cognitive behavioral psychotherapist, Rakitzi, Stavroula
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAKITZI & GEORGILA CBT
Record Dates: First submitted 2025-04-23; First posted 2025-05-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Anxiety; Depression; Obsessive-compulsive Disorder; Personality Disorder; Bipolar Disorder; Schizophrenia; Psychotic Disorders; PTSD
Keywords: Pharmacotherapy; Cognitive behavioral psychotherapy; Recovery
MeSH Terms: conditions — Anxiety Disorders; Depression; Obsessive-Compulsive Disorder; Personality Disorders; Bipolar Disorder; Schizophrenia; Psychotic Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Group A (Experimental): The combination of pharmacotherapy (anxiolytics (Tavor, clonotril, lexotanil), antidepressants (SSRI, SNRI)) and individual cognitive behavioral psychotherapy by anxiety disorders and depression.
  20 patients
  Interventions: Combination Product: Group A. The combination of pharmacotherapy and individual cognitive behavioral psychotherapy by anxiety disorders and depression.
- Group B (Experimental): The combination of pharmacotherapy (anxiolytics (Tavor, clonotril, lexotanil), antidepressants (SSRI, SNRI)) and individual cognitive behavioral psychotherapy by PTSD.
  12 patients
  Interventions: Combination Product: Group B. The combination of pharmacotherapy and individual cognitive behavioral psychotherapy by PTSD
- Group C (Experimental): The combination of pharmacotherapy (anxiolytics (Tavor, clonotril, lexotanil), antidepressants (SSRI, SNRI)) and individual cognitive behavioral psychotherapy by obsessive-compulsive disorder.
  15 patients
  Interventions: Combination Product: Group C. The combination of pharmacotherapy and individual cognitive behavioral psychotherapy by obsessive-compulsive disorder.
- Group D (Experimental): The combination of pharmacotherapy (anxiolytics ((Tavor, clonotril, lexotanil), antidperessants (SSRI, SNRI), mood stabilizers (Lithium, depakine) and antipsychotics (clozapine and atypical antipsychotics)) and individual cognitive behavioral psychotherapy by bipolar disorders.
  15 patients
  Interventions: Combination Product: Group D.The combination of pharmacotherapy and individual cognitive behavioral psychotherapy by bipolar disorder
- Group E (Experimental): The combination of pharmacotherapy (antipsychotics (clozapine and atypical antipsychotics)) , anxiolytics (Tavor, clonotril, lexotanil), antidepressants (SSRI, SNRI)) and individual cognitive behavioral psychotherapy by schizophrenia and psychotic disorders.
  20 patients
  Interventions: Combination Product: Group E. The combination of pharmacotherapy and individual cognitive behavioral psychotherapy by schizophrenia and psychotic disorders
- Group F (Experimental): The combination of pharmacotherapy (antidepressants (SSRI, SNRI), anxiolytics (Tavor, clonotril, lexotanil) antipsychotics (clozapine and atypical antipsychotics)) and individual cognitive behavioral psychotherapy by personality disorders.
  20 patients (2 narcistic personality disorder, 5 borderline personality disorder, 4 obsessive-compulsive disorder, 5 avoidant personality disorder, 4 depedent personality disorder)
  Interventions: Combination Product: Group F.The combination of pharmacotherapy and individual cognitive behavioral psychotherapy by personality disorders

INTERVENTIONS:
Combination Product: Group A. The combination of pharmacotherapy and individual cognitive behavioral psychotherapy by anxiety disorders and depression. — The combination of pharmacotherapy (anxiolytics (tavor, clonotril, lexotanil), antidepressants (SSRI, SNRI) and individual cognitive behavioral psychotherapy by anxiety disorders and depression.
  Arms: Group A
Combination Product: Group B. The combination of pharmacotherapy and individual cognitive behavioral psychotherapy by PTSD — The combination of pharmacotherapy (anxiolytics (tavor, clonotril, lexotanil), antidepressants (SSRI, SNRI) and individual cognitive behavioral psychotherapy by PTSD
  Arms: Group B
Combination Product: Group C. The combination of pharmacotherapy and individual cognitive behavioral psychotherapy by obsessive-compulsive disorder. — The combination of pharmacotherapy and individual cognitive behavioral psychotherapy by obsessive-compulsive disorder.
  Arms: Group C
Combination Product: Group D.The combination of pharmacotherapy and individual cognitive behavioral psychotherapy by bipolar disorder — The combination of pharmacotherapy (anxiolytics (tavor, clonotril, lexotanil) antidepressants (SSRI, SNRI), mood stabilizers (lithium, depakine), antipsychotics (clozapine and atypical antipsychotics)) and individual cognitive behavioral psychotherapy by bipolar disorder.
  Arms: Group D
Combination Product: Group E. The combination of pharmacotherapy and individual cognitive behavioral psychotherapy by schizophrenia and psychotic disorders — The combination of pharmacotherapy (anxiolytics(tavor, clonotril, lexotanil), antidepressants (SSRI, SNRI), antipsychotics (clozapine and atypical antipsychotics)) and individual cognitive behavioral psychotherapy by schizophrenia and psychotic disorders.
  Arms: Group E
Combination Product: Group F.The combination of pharmacotherapy and individual cognitive behavioral psychotherapy by personality disorders — The combination of pharmacotherapy (anxiolytics (tavor, clonotril, lexotanil), antidepressants (SSRI, SNRI), antipsychotics (clozapine and atypical antipsychotics) and individual cognitive behavioral psychotherapy by personality disorders.
  Arms: Group F

SUMMARY:
The combination of pharmacotherapy and individual cognitive behavioral therapy in a private practice.

DETAILED DESCRIPTION:
Reintegration into society and good functional outcome by people with mental health disorders is frequently the result of the combination of pharmacotherapy and individual cognitive behavioral psychotherapy. The effectiveness and efficacy of this combination of treatments under the recovery perspective by anxiety disorders, depressive disorders, PTSD, bipolar disorders, schizophrenia and psychotic disorders, by obsessive-compulsive disorders and by personality disorders presents the main goal of this research protocol. Recovery means that people learn through the trherapy to be responsible towards their own problems.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65,
* IQ ≥ 80,
* Diagnosis: anxiety disorders, depression, obsessive-compulsive disorders, PTSD, personality disorders, bipolar disorders, schizophrenia and psychotic disorders.

Exclusion Criteria:

*Substance abuse and head injury.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2025-06-02 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
MCCB BACS symbol coding | Preintervention
  It measures speed of processing. Minimum 0, maximum 110, high scores better
MCCB BACS symbol coding | Immediately after the intervention
  It measures speed of processing. Minimum 0, maximum 110, high scores better
MCCB BACS symbol coding | Follow-up up to 24 weeks
  It measures speed of processing. Minimum 0, maximum 110, high scores better
MCCB Wechsler memory scale-spatial span | Preintervention
  It measures non-verbal working memory. Minimum 0, maximum 32, high scores better, Summary of forward and backward total score.
MCCB Wechsler memory scale-spatial span | Immediately after the intervention
  It measures non-verbal working memory. Minimum 0, maximum 32, high scores better, Summary of forward and backward total score.
MCCB Wechsler memory scale-spatial span | Follow-up up to 24 weeks
  It measures non-verbal working memory. Minimum 0, maximum 32, high scores better, Summary of forward and backward total score.
MCCB Neurospychological Assessment Battery (NAB) | Preintervention
  It measures reasoning and problem-solving. Minimum 0, maximum 26. high scores better
MCCB Neurospychological Assessment Battery (NAB) | Immediately after the intervention
  It measures reasoning and problem-solving. Minimum 0, maximum 26. high scores better
MCCB Neurospychological Assessment Battery (NAB) | Follow-up up to 24 weeks
  It measures reasoning and problem-solving. Minimum 0, maximum 26. high scores better
MCCB Brief visuospatial memory test | Preintervention
  It measures visual memory. Sum of Trial 1, 2, 3. Minimum 0, maximum 12. high scores better
MCCB Brief visuospatial memory test | Immediately after the intervention
  It measures visual memory. Sum of Trial 1, 2, 3. Minimum 0, maximum 12. high scores better
MCCB Brief visuospatial memory test | Follow-up up to 24 weeks
  It measures visual memory. Sum of Trial 1, 2, 3. Minimum 0, maximum 12. high scores better
The Greek verbal memory test | Preintervention
  It measures oral verbal memory. Semantic. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better.
The Greek verbal memory test | Immediately after the intervention
  It measures oral verbal memory. Semantic. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better.
The Greek verbal memory test | Follow-up up to 24 weeks
  It measures oral verbal memory. Semantic. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better.
The Greek verbal memory test | Preintervention
  It measures oral verbal memory. Semantic. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better
The Greek verbal memory test | Immediately after the intervention
  It measures oral verbal memory. Semantic. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better
The Greek verbal memory test | Follow-up up to 24 weeks
  It measures oral verbal memory. Semantic. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better
The Greek verbal memory test | Preintervention
  It measures oral verbal memory. Phonological. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better
The Greek verbal memory test | Immediately after the intervention
  It measures oral verbal memory. Phonological. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better
The Greek verbal memory test | Follow-up up to 24 weeks
  It measures oral verbal memory. Phonological. Sum of the 3 categories divided to 3. Minimum 0, maximum 40. high scores better
The Greek verbal memory test | Preintervention
  It measures written verbal memory. Sum of the 2 tasks. Minimum 0, maximum as much as possible. high scores better.
The Greek verbal memory test | Immediately after the intervention
  It measures written verbal memory. Sum of the 2 tasks. Minimum 0, maximum as much as possible. high scores better.
The Greek verbal memory test | Follow-up up to 24 weeks
  It measures written verbal memory. Sum of the 2 tasks. Minimum 0, maximum as much as possible. high scores better.
SCL-90-R | Preintervention
  It evaluates psychopathology. T>60 means psychopathology. Low scores better
SCL-90-R | Immediately after the intervention
  It evaluates psychopathology. T>60 means psychopathology. Low scores better
SCL-90-R | Follow-up up to 24 weeks
  It evaluates psychopathology. T>60 means psychopathology. Low scores better
PANNS total | Preintervention
  It measures positive, negative symptoms and general psychopathology. Minimum 31, maximum 210. Low scores better
PANNS total | Immediately after the intervention
  It measures positive, negative symptoms and general psychopathology. Minimum 31, maximum 210. Low scores better
PANNS total | Follow-up up to 24 weeks
  It measures positive, negative symptoms and general psychopathology. Minimum 31, maximum 210. Low scores better
WHODAS total | Preintervention
  It measures functional outcome. Minimum 0, maximum 100. low scores better.
WHODAS total | Immediately after the intervention
  It measures functional outcome. Minimum 0, maximum 100. low scores better.
WHODAS total | Follow-up up to 24 weeks
  It measures functional outcome. Minimum 0, maximum 100. low scores better.
RAS-DS total | Preintervention
  It measures recovery. Minimum 0, maximum 152. High scores better.
RAS-DS total | Immediately after the intervention
  It measures recovery. Minimum 0, maximum 152. High scores better.
RAS-DS total | Follow-up up to 24 weeks
  It measures recovery. Minimum 0, maximum 152. High scores better.
The Clinical Global Impression Scale (CGI) | Preintervention
  It measures severity of illness. Minimum 0, Maximum 7, low scores better.
The Clinical Global Impression Scale (CGI) | Immediately after the intervention
  It measures severity of illness. Minimum 0, Maximum 7, low scores better.
The Clinical Global Impression Scale (CGI) | Follow-up up to 24 weeks
  It measures severity of illness. Minimum 0, Maximum 7, low scores better.
The Clinical Global Impression Scale (CGI) | Preintervention
  It measures global improvement. Minimum 0, Maximum 7, low scores better.
The Clinical Global Impression Scale (CGI) | Immediately after the intervention
  It measures global improvement. Minimum 0, Maximum 7, low scores better.
The Clinical Global Impression Scale (CGI) | Follow-up up to 24 weeks
  It measures global improvement. Minimum 0, Maximum 7, low scores better.
SRSDA | Preintervention
  It measures Depression. Minimum 0, maximum 14 or higher. Low scores better
SRSDA | Immediately after the intervention
  It measures Depression. Minimum 0, maximum 14 or higher. Low scores better
SRSDA | Follow-up up to 24 weeks
  It measures Depression. Minimum 0, maximum 14 or higher. Low scores better
SRSDA B | Preintervention
  It measures Anxiety. Minimum 0, maximum 10 or higher. Low scores better
SRSDA B | Immediately after the intervention
  It measures Anxiety. Minimum 0, maximum 10 or higher. Low scores better
SRSDA B | Follow-up up to 24 weeks
  It measures Anxiety. Minimum 0, maximum 10 or higher. Low scores better
Hamilton Depression Scale | Preintervention
  It measures depression. Minimum 0, maximum 23. Low scores better.
Hamilton Depression Scale | Immediately after the intervention
  It measures depression. Minimum 0, maximum 23. Low scores better.
Hamilton Depression Scale | Follow-up up to 24 weeks
  It measures depression. Minimum 0, maximum 23. Low scores better.
Montgomery and Asperg depression scale | Preintervention
  It measures depression. Minimum 0, maximum 60. Low scores better.
Montgomery and Asperg depression scale | Immediately after the intervention
  It measures depression. Minimum 0, maximum 60. Low scores better.
Montgomery and Asperg depression scale | Follow-up up to 24 weeks
  It measures depression. Minimum 0, maximum 60. Low scores better.
The Altman self-rating scale | Preintervention
  It measures mania. Minimum 0, maximum 6 or higher. Low scores better.
The Altman self-rating scale | Immediately after the intervention
  It measures mania. Minimum 0, maximum 6 or higher. Low scores better.
The Altman self-rating scale | Follow-up up to 24 weeks
  It measures mania. Minimum 0, maximum 6 or higher. Low scores better.
The Young mania rating scale | Preintervention
  It measures mania. Minimum 0, maximum 60. Low scores better
The Young mania rating scale | Immediately after the intervention
  It measures mania. Minimum 0, maximum 60. Low scores better
The Young mania rating scale | Follow-up up to 24 weeks
  It measures mania. Minimum 0, maximum 60. Low scores better
PSYRAT H | Preintervention
  It measures psychotic symptoms. Hallucinations. Minimum 0, maximum 24. Low scores better.
PSYRAT H | Immediately after the intervention
  It measures psychotic symptoms. Hallucinations. Minimum 0, maximum 24. Low scores better.
PSYRAT H | Follow-up up to 24 weeks
  It measures psychotic symptoms. Hallucinations. Minimum 0, maximum 24. Low scores better.
PSYRAT D | Preintervention
  It measures psychotic symptoms. Delusions. Minimum 0, maximum 44. Low scores better
PSYRAT D | Immediately after the intervention
  It measures psychotic symptoms. Delusions. Minimum 0, maximum 44. Low scores better
PSYRAT D | Follow-up up to 24 weeks
  It measures psychotic symptoms. Delusions. Minimum 0, maximum 44. Low scores better

SECONDARY OUTCOMES:
WAIS | Preintervention
  It measures the Intelligenz-quotient. For bipolar disorder, schizophrenia and psychotic disorders

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Stavroula Rakitzi, PhD, Study Director — Private Practice; Dr. Polyxeni Georgila, M. D., Study Director — Private Practice
Locations (1):
- Private practice of Dr. S. Rakitzi and Dr. P. Georgila ILISION 34 15771 ATHENS GREECE, Athens, Greece

IPD SHARING:
Plan to Share IPD: No
This is our first effectiveness study regarding pharmacotherapy and cognitive behavioral psychotherapy in our private practice.

REFERENCES:
- [Background] 2. Aster, M., Neubauer, M., & Horn R. (2006) Wechsler-Intelligenztest für Erwachsene WIE. Frankfurt: Harcourt Test Services.
- [Background] Altman EG, Hedeker D, Peterson JL, Davis JM. The Altman Self-Rating Mania Scale. Biol Psychiatry. 1997 Nov 15;42(10):948-55. doi: 10.1016/S0006-3223(96)00548-3. PMID 9359982
- [Background] Bech, P. (1993). Rating scales for Psychopathology, Health Status and Quality of Life. Berlin, Heidelberg, New York: Springer-Verlag.
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Donias, S., Karastergiou, A., & Manos N. (1991). Standardization of the symptom checklist-90-R rating scale in a Greek population. Psychiatriki, 2(1), 42-48
- [Background] Fountoulakis KN, Iacovides A, Kleanthous S, Samolis S, Gougoulias K, St Kaprinis G, Bech P. The Greek translation of the symptoms rating scale for depression and anxiety: preliminary results of the validation study. BMC Psychiatry. 2003 Dec 10;3:21. doi: 10.1186/1471-244X-3-21. PMID 14667249
- [Background] Guy, W. (ed). (1976). ECDEU Assessment. Manual for Psychopharmacology. Rockville, MD: US Department of Heath, Education, and Welfare Public Health Service Alcohol, Drug Abuse, and Mental Health Administration, 1976
- [Background] Haddock G, McCarron J, Tarrier N, Faragher EB. Scales to measure dimensions of hallucinations and delusions: the psychotic symptom rating scales (PSYRATS). Psychol Med. 1999 Jul;29(4):879-89. doi: 10.1017/s0033291799008661. PMID 10473315
- [Background] Hancock, N., Scanlan, J.N., Bundy, A.C., Honey, A. (2019). Recovery Assessment Scale -Domains & Stages (RAS-DS) Manual- Version 3. Sydney: University of Sydney.
- [Background] Hancock, N., & the University of Sydney (2023). Rakitzi S. Katoudi S. Recovery Assessment Scale-Domains & Stages (RAS-DS). The Greek version.
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] .Kosmidou, M., & Vlahou, Ch. (2010). The Greek verbal memory test. Athens: Parisianos.
- [Background] Koumpouros, Y., Papageorgiou, E., & Sakellari E. et al. (2018). Adaptation and psychometric properties evaluation of the Greek version of WHODAS 2.0. Pilot application in Greek elderly population. Health Services and Outcomes Research Methodology, 18(1), 63-74. https://doi.org/10.1007/s10742-017- 0176-x
- [Background] .Lykouras, L., Botsis, A., & Oulis P. (2005). The PANSS Scale. Athens: Scientific Publications
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Rakitzi, S. (2023). Clinical psychology and cognitive behavioral psychotherapy. Recovery in mental health. Springer
- [Background] Williams JB, Kobak KA. Development and reliability of a structured interview guide for the Montgomery Asberg Depression Rating Scale (SIGMA). Br J Psychiatry. 2008 Jan;192(1):52-8. doi: 10.1192/bjp.bp.106.032532. PMID 18174510
- [Background] World Health Organization. International classification of functioning, disability and health (ICF). Geneva: World Health Organization; 2001
- [Background] Young RC, Biggs JT, Ziegler VE, Meyer DA. A rating scale for mania: reliability, validity and sensitivity. Br J Psychiatry. 1978 Nov;133:429-35. doi: 10.1192/bjp.133.5.429. PMID 728692

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT06993662/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT06993662/ICF_001.pdf